CLINICAL TRIAL: NCT05217108
Title: A Mobile Phone Text-based Intervention to Reduce Sedentary Behavior and Engage Communities on the Importance of Healthy Lifestyles: the TEXT2MOVE Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-1014; NCI-2022-00101 (Other: NCI CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-01-05; First posted 2022-02-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Life Style; Healthy Lifestyle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fit Bit (Study Groups) (Other): Participants wear a Fitbit every day for 8 weeks to record the number of steps you take
  Interventions: Device: FitBit

INTERVENTIONS:
Device: FitBit — All participants in each study group will receive a Fitbit. Participants will be asked to wear a Fitbit every day for 8 weeks to record the number of steps you take

SUMMARY:
To learn if an 8-week, phone-based texting intervention program will reduce sedentary (non-mobile) behavior.

DETAILED DESCRIPTION:
Primary Objective: To test the effect of two text messaging strategies, responsive texts and standard scheduled texts, on sedentary behavior in a racially and geographically diverse sample of adults.

Secondary Objective: To assess participant engagement with the program and with the educational content delivered via text messaging.

Exploratory Objective: To determine whether two text messaging strategies, responsive texts and standard scheduled texts, increases physical activity in a racially and geographically diverse sample of adults.

Exploratory Objective: To determine whether two text messaging strategies, responsive texts and standard scheduled texts are associated with changes in corresponding patient attitudes as assessed by surveys of exploring sedentary behavior, readiness for exercise change, and physical functioning.

ELIGIBILITY:
Inclusion criteria:

1. >18 years old
2. owns a smart phone
3. has access to WiFi or willing to use mobile data
4. has an email address or willing to create an email address
5. able to read and understand English;
6. able to give informed consent;
7. willing to receive text messages and complete brief questionnaires on their smart phone
8. self-reports sedentary behavior (> 6 hours/day of sitting time).

Exclusion criteria:

1. unwilling to have sedentary behavior and activity tracked
2. unable to walk without ambulatory assistance device (i.e. cane or walker) or due to underlying medical condition
3. MD Anderson employees that report to the Principal Investigators of this study
4. family or household member already enrolled into study
5. not sedentary based on < 6 hours/day of sitting time, and (6) currently participating in a weight management or exercise study or program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Daily minutes in sedentary behavior based on Fitbit data. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org